CLINICAL TRIAL: NCT01285882
Title: Representations of Transplantation in Patients With Mucoviscidosis, in Their Assistants and in Their Medical Persons
Brief Title: Representations of Transplantation in Patients and in Health Care Professionals
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Anne OMNES, Nantes University Hospital
Other Study IDs: PROG/10/89
Record Dates: First submitted 2011-01-27; First posted 2011-01-28 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Cystic Fibrosis
Keywords: Lung transplantations; Representations; Mucoviscidosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Artificial Intelligence

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Representations
  Interventions: Other: Representations

INTERVENTIONS:
Other: Representations — 1. A pre-test with 5 medical persons and 5 persons without mucoviscidosis will be realized to adjust the tools and place of the interview.
  2. To collect analyzable data for 30 patients, 40 patients will be included in the study. A conceptual card will be associated to a semi-structured interviews to gather information.Two subgroups will be considered in th a analysis :
     * 1st sub-group : After the announcement of the transplant indication by the doctor and before the consultation in the transplant centre.
     * 2nd subgroup : After the consultation in the transplant centre but before the inscription on the waiting list. The analysis of conceptual cards in these two subgroups will permit to study the differences between the representations of patients before and after the consultation in the transplant centre.
  3. Realize a 2nd interview on the same principle with all patients, 1 year after their lung transplantation.

SUMMARY:
Main objective : This project aims to have a better understanding of the influence of representations of patients with mucoviscidosis, their assistants and their medical persons in the choice of patients to accept or not lung transplantation.

Specific objectives :

1. Identify the knowledge, representations, or feelings of patients which could constitute bridles or factors of motivation to use for transplantation.
2. Identify the knowledge, representations, or feelings of medical persons which could constitute bridles or factors of motivation to the "encouraging" proposal to patients of lung transplant.
3. Identify the knowledge, representations, or feelings of assistants which could constitute bridles or factors of motivation to the "encouragement" of lung transplantation at its close.
4. Identify the needs of patients, assistants and medical persons to successfully reduce these bridles to transplantation and increase the factors of motivation.
5. Compare the representations of patients, assistants and medical persons
6. Search representations associated with patients who refuse the transplantation and those who accept the transplantation

ELIGIBILITY:
Inclusion Criteria:

* For patients :

  * Adult patient (those concerned by the suggestion of lung transplant).
  * At the time of transplant indication : after the first suggestion of the medical person, before or after the preoperative graft check-up but before registration on waiting list.
* For medical persons :

  * Medical persons involved in the suggestion of lung transplantation to the patients.
* For assistants :

  * Adult close to the patient and that the patient sees as a resource person and advisor in his choices for the transplant : reference person having a major influence for the patient (spouse, parent, sibling, friend ...)

Exclusion Criteria:

* For patients :

  * Patient with a psychiatric disorder
  * Patient in intensive care unit
  * Palliative care patient
  * Patient aged under 18 years old
  * Patient refusal
* For medical persons :

  * Medical person refusal
* For assistants :

  * Assistant or patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients for whom a lung transplant indication is established
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie DAVID, Doctor, Principal Investigator — Nantes University Hospital; Raphaële NOVE-JOSSERAND, Doctor, Study Chair — Hospices Civils de Lyon; Marc STERN, Profesor, Study Chair — Hôpital Foch; Martine REYNAUD-GAUBERT, Profesor, Study Chair — CHU de Marseille; Isabelle DURIEU, Doctor, Study Chair — Hospices Civils de Lyon; Dominique HUBERT, Doctor, Study Chair — Hôpital Cochin; Sophie RAMEL, Doctor, Study Chair — Centre de Perharidy - Roscoff; RAVONINJATOVO, Doctor, Study Chair — CHU de Reims; Magali DUPUY-GRASSET, Doctor, Study Chair — University Hospital, Limoges; Céline MENETREY, Doctor, Study Chair — University Hospital, Limoges; Chantal BELLEGUIC, Doctor, Study Chair — Rennes University Hospital; Corina SANZIANA CORHUT, Doctor, Study Chair — Central Hospital, Nancy, France; Benoît GODBERT, Doctor, Study Chair — Central Hospital, Nancy, France; Françoise VARAIGNE, Doctor, Study Chair — CHU de Tours; Isabelle PIN, Doctor, Study Chair — University Hospital, Grenoble; Marie-Laure UFFREDI, Doctor, Study Chair — CH de Vannes
Locations (1):
- Nantes University Hospital, Nantes, France